CLINICAL TRIAL: NCT05391295
Title: Mapping Emotional Dynamics in Cutaneous T-cell Lymphoma (Type Mycosis Fungoides and/or Sezary Syndrome) Patients and Chronic Cluster Headache Patients During Treatment With Corticosteroids: a Case Series Study
Brief Title: Mapping Emotional Dynamics During Corticosteroid Treatment
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Erik J. Giltay, MD, PhD, Principal Investigator, Leiden University Medical Center
Other Study IDs: W2022.002
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Emotions; Corticosteroids

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 6 CTCL patients, and 6 chronic cluster headache patients: The patients will be treated according to standard regular care, which is a corticosteroid treatment regime.
  Interventions: Other: Short daily questionnaire

INTERVENTIONS:
Other: Short daily questionnaire — This study includes 1 survey that needs to be filled out by the patient on his/her phone daily during the course of corticosteroid treatment. The investigators will start the survey few days before the corticosteroid treatment and it will continue till the end of the treatment regime. The treatment regime is regular care and patient specific, but will approximately have a duration of 40 days. In case of prolonged treatment with steroids it is decided to have a limit for our study: either until 7 days after the end of corticosteroid treatment or a maximum of 60 days.

SUMMARY:
Rationale: Synthetic glucocorticoids can result in neuropsychiatric adverse effects in a minority of patients. Although, not all patients experience severe adverse effects, more subtle emotional disturbances are often experienced. With a variation on ecological momentary assessment (EMA), with a daily assessment, the investigators will collect the patient's emotional symptoms in real time and in the patients natural environment during corticosteroid treatment. With dynamic time warping (DTW) analysis the investigators aim to analyse the temporal dynamics of different emotional states and visualize these emotional dynamics over time. The patient dermatologist and neurologist will receive the idiographic results as a feedback form, which may give insights into temporal (and possibly causal) central emotions, which may help to overcome mood disturbances.

Objective: Mapping emotional dynamics with DTW analysis in 6 mycosis fungoides or Sezary syndrome patients and 6 chronic cluster headache patients treated with systemic corticosteroids.

Study design: Case series report study. Study population: Six patients with cutaneous T-cell lymphoma (type mycosis fungoides and/or Sezary syndrome), and six patients with cluster headache.

Main study parameters/endpoints: An idiographic DTW analysis of emotional dynamics during and after corticosteroid treatment in six mycosis fungoides and/or Sezary syndrome patients, and six chronic cluster headache patients.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no additional risks associated with study participation. The patients who will participate in this case series study need to complete a 5-minute survey daily using a m-Path smartphone app during corticosteroid treatment. The data analysis may increase the insight into centrality measures of emotions and the emotional clusters for the individual patient.

DETAILED DESCRIPTION:
This is a case series study in which we want to map emotional dynamics with DTW analysis in 6 mycosis fungoides and/or Sezary syndrome patients and 6 chronic cluster headache patients, who will be treated with a corticosteroid regime. Duration of the study will approximately be 40-60 days, depending on the duration of the treatment:

* The mycosis fungoides and/or Sezary syndrome patients are treated for approximately 40 days.
* The chronic cluster headache patients are treated for approximately 60 days.

The patient will be treated according to standard regular care. This will not change. For study purposes, a 15 minute explanation of the survey will be given. We will ask the patient to install the m-Path app on their smartphone, and to complete the daily survey (with 23 statements with a slider) on his/her phone during the treatment period, which will take approximately 5 minutes per day. At the end of the study the patient will get the results visualized, with a 30 minute explanation of the results, which may increase insights of the patient's emotions dynamics over time during corticosteroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Mycosis fungoides and/or Sezary syndrome patients
* Chronic cluster headache patients
* Corticosteroid treatment

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mycosis fungoides and/or Sezary syndrome patients and cluster headache patients who will be treated according to standard regular care, which is a corticosteroid treatment regime.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Mapping emotional dynamics with DTW analysis in CTCL patients and cluster headache patients treated with corticosteroids. | Short daily questionnaire for +- 1 month or +- 2 months
  A dynamic time warping (DTW) analysis on the data.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Giltay, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- LUMC, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided